CLINICAL TRIAL: NCT04180293
Title: Family Psychoeducation for Military Veterans: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Abraham Rudnick, Clinical Director, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18200
Record Dates: First submitted 2019-11-13; First posted 2019-11-27 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Veterans Family; Military Family; Trauma, Psychological
Keywords: Military; Veteran; Family; Psychoeducation; Resiliency; Operational stress injuries; Post traumatic stress disorder
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic | interventions — Program Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Military Veterans and their families (Other): This group will participate in both the pilot psychoeducation program and its evaluation.
  Interventions: Behavioral: Pilot psychoeducation program; Other: Program evaluation

INTERVENTIONS:
Behavioral: Pilot psychoeducation program — Canadian Armed Forces veterans and their family members will be recruited to participate in this pilot virtual psychoeducation program and its evaluation. Two six-week sessions will be implemented over a virtual care platform (Zoom for healthcare) based out of OSI Clinic in Atlantic Canada - the first in January/February of 2021 and the second in the spring of 2021. A maximum of 10-15 participants (including both veterans and their family members) will be recruited for each group. Family members are defined as spouses/partners, siblings, parents, and adult children. Each of the weekly sessions will take place virtually and will be led by at least two trained facilitators (one from the research team, and one member of the OSI clinical staff team). Each of these sessions will focus on providing education of different topics relevant to those accessing services at the clinic (e.g., types of treatments available, tools to support families, self care, etc.).
Other: Program evaluation — At the end of each six-week session, program outcomes will be assessed qualitatively by a member of the research team. Participants will take part in semi-structured interviews guided by questions informed by the ecological family systems theory.

SUMMARY:
Operational Stress Injuries (OSIs), including post traumatic stress disorder (PTSD), are prevalent among veterans deployed in recent combat missions, the effects of which are experienced within their families. The development of evidence-based programs for veterans with OSIs and their families is critical because family functioning both affects and is affected by OSIs. Few programs have been implemented, however, particularly in Canada, and those that have are not evaluated. Research suggests that brief, systems-focused family psychoeducation programs are useful in the treatment of OSIs, specifically PTSD, leading to increases in targeted PTSD knowledge and skills and enhancing resilience.

The purpose of this pilot study is to: (1) develop a systems-focused, virtual psychoeducational program designed to enhance resilience in veterans with OSIs receiving clinical care at an OSI clinic in Atlantic Canada and their families; (2) to implement the virtual program with veterans and their families at the OSI clinic; (3) to evaluate the efficacy of the program; and (4) to compare resilience-building family psychoeducation to the standard information-providing services currently available to families at the OSI clinic. Results will be shared within the network of OSI clinics in Canada and will inform the development of a proposal for a mixed-method study.

DETAILED DESCRIPTION:
Context

The capacity of military and veteran families to develop and maintain positive mental health and well-being is challenged by contemporary operational imperatives. Since 1990, the Canadian Armed Forces (CAF) has engaged in more than 20 major international operations, involving multiple rotations of members serving in complex missions including Rwanda, Bosnia, Afghanistan, and, more recently, Mali. The intensified operational tempo is associated with an increase in the prevalence of operational stress injuries (OSIs). OSIs are persistent psychological difficulties resulting from operational duties performed while serving in the CAF. OSIs span a spectrum, including diagnosed psychiatric conditions such as anxiety disorders, depression, and post-traumatic stress disorder (PTSD) as well as other conditions that may be less severe, but still interfere with daily functioning. In a recent iteration of the Life After Service Study (LASS), a national survey of CAF veterans receiving services from Veterans Affairs Canada (VAC), 23% reported a diagnosis of one or more mental disorders, 5.8% reported suicidal ideation, and 1.1% reported a suicide attempt in the previous year. Specialized OSI clinics are now in place to support treatment-seeking veterans who qualify for care through VAC. An increase in mental health diagnoses requiring clinical management in these clinics has been documented.

The effects of OSIs in members and veterans ripple through their families. Results of a recent study focusing on the impacts of OSIs on the mental health and well-being of families of CAF veterans suggest that the imperative to care for the veteran becomes the central, organizing facet of family experience. In response, family structure, including family role redefinition and reallocation, shifts. Spouses assume full responsibility for family functioning and adapt routines, as required, while providing care to the veteran. Some spouses describe themselves as caregivers to the veteran, performing daily work that involves mediating and buffering the internal and external stresses affecting him/her. Consequently, spouses report burn out and specific health conditions attributed to the stress emerge. These health outcomes develop in an environment characterized by loss of identity and social and geographic isolation for some. Emotional stress, relationship tensions, and financial concerns resulting from changes in employment impact the whole family. Throughout, family members must reconcile the loss of the veteran as he/she once was. In some cases, children share these burdens, enacting role behavior incompatible with their developmental stage. Children may also experience emotional and behavioural problems.

Some veteran families cope with these challenges successfully, developing resilience through practical task management, problem-solving, and social support. Family resilience results from the interplay of individual assets and the social contexts in which they develop. Maintaining shared family beliefs, facilitating family organization, and communicating are processes that facilitate resilience through stress and adversity. Maintaining shared beliefs helps family members make sense of stress and adversity. Shared beliefs can be introduced or reintroduced to the family system through religious, spiritual practice, artistic expression, or through connection with family rituals or the natural environment. Furthermore, some research suggests that agency and self-determination are mobilized through shared belief systems and are instrumental in efforts to reinterpret adversity as a challenge that can be mastered.

Family organization enables families to manage the impacts of OSIs on both the veteran and the family system. Clear and consistent organizational patterns reassure family members, particularly vulnerable family members such as children, that, notwithstanding the adversity and stress, the structure of the family is continuous, dependable, and strong.

Communication processes are also important in resilient families. Clear and unambiguous messages, empathetically and openly shared, encourage inclusion, collaborative problem-solving, and conflict resolution.

For families experiencing adversity, such as the stresses associated with supporting a veteran living with an OSI, resilience processes enable families to recover or "bounce back" by developing "resistance to psychosocial risk experiences" or to reconfigure by "bouncing forward" as new capacities are developed. Resilience is not innate or merely a function of individual personality traits. Rather, it can be learned and developed.

Brief, systems-focused psychoeducational programs have the potential to support the development of veteran family resilience. These programs enhance individual and relational capacities that reduce psychological and relational distress. The tools required to navigate interconnected systems (informal and formal social networks) can also be acquired. Early identification of issues and enhancement of help-seeking behaviours are the focus of psychoeducational programs. They are a complement to therapy, not a replacement. Indeed, brief, systems-focused programs attract and retain families in need who are unlikely to seek out therapeutic intervention and have a significant role to play in addressing their complex needs.

To date, evidence-based, psychoeducational programs for veterans with OSIs and their families are few in number, particularly in Canada. Some research is ongoing in the United States. For example, the efficacy of psychoeducation for veterans with OSIs and their families was measured in an American study involving 100 veterans with PTSD and 96 family members participating in a longitudinal evaluation of a program entitled REACH (Reaching out to Educate and Assist Caring, Healthy Families). Results indicate that participation in REACH positively impacts both veterans with PTSD and their family members. Participants showed improvements in knowledge about PTSD, family adaptation strategies, family communication, and empowerment. Relationship satisfaction, perceived social support, and a decrease in PTSD symptoms were also reported.

The purpose of this pilot study is to contribute to the development of evidence-based, systems-focused virtual psychoeducational programming for CAF veterans with OSIs and their families. This initiative will draw upon partnerships and expertise at an OSI Clinic in Atlantic Canada.

Theoretical Framework

This pilot program will be developed as a brief, systems-focused virtually-delivered psychoeducational program. Therefore, the ecological family systems theory will serve as a foundation for the development of the content of the pilot program and its evaluation. Grounded in a bioecological model of human development, the original ecological family systems model and its subsequent iterations bring into view a system of four interconnected environments (microsystem, mesosystem, exosystem, and macrosystem), each representing the interdependent contexts embodied in the lives of individuals and families. These environments and their roles in developing and maintaining resilience will constitute program components. For example, loss of identity, shared beliefs, role redefinition/reallocation (microsystem), changes in routines, caregiving imperatives, family organization strategies (mesosystem), military and veteran family policies (exosystem), and military culture (macrosystem) and the processes integral to navigating these interconnected systems will be explored. The non-normative changes in roles and environments, or the ecological transitions, particular to the military context that challenge resilience for the families of veterans with OSIs will also be considered.

Methodology

CCAF veterans diagnosed with an OSI at least one year prior to the start of the study and receiving care through the OSI Clinic in Dartmouth, N.S. and their family members will be recruited to participate in the pilot program and its evaluation. Two six-week virtual sessions will be implemented at the clinic - the first in January/February of 2021 and the second in the spring of 2021. A maximum of 10-15 participants (including both veterans and their family members) will be recruited for each group. Family members are defined as spouses/partners, siblings, parents, and adult children. Prior to the start of the program, participants will be qualitatively interviewed by a member of the research team. Participants will take part in interviews guided by questions informed by the ecological family systems theory. Program participants will be interviewed using a semi-structured interview guide; see interview guide included in attached appendices. Interviews will be taped and transcribed verbatim. Field notes identifying observations, thoughts, and additional information contributing to the formative analysis of the data will be maintained.

Each of the weekly sessions will take place over a virtual care platform (Zoom for Healthcare) and will be led by at least two trained facilitators (one from the research team, and one member of the OSI clinical staff team). Each of these sessions will focus on providing education of different topics relevant to those accessing services at the clinic (e.g., types of treatments available, tools to support families, self care). See attached appendix for draft outline of group sessions. The facilitators will also be there to support the participants with any questions they may have. The OSI clinical team member facilitating these groups will also be able to meet individually with the client outside of the group as needed to provide additional support.

At the end of each six-week session, program outcomes will be assessed qualitatively by a member of the research team utilizing the same interview guide as mentioned above. Six weeks after the end of the session, participants will be interviewed again as a final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Canadian Armed Forces (CAF) veterans who wish to participate in this study must be:

  1. Living with a diagnosed Operational Stress Injury (OSI) for at least one year prior to the start of the study.
  2. Receiving care at the OSI Clinic in Dartmouth.
* Family members who wish to participate may include:

  1. Spouses/partners;
  2. Siblings;
  3. Parents;
  4. Adult children (older than 19 years of age).

Exclusion Criteria:

* Active serving members of the CAF.
* Active and former members of the Royal Canadian Mounted Police.
* Children (younger than 19 years of age).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Patient and family-perceived efficacy and utility of a pilot psychoeducation program. | Final Interviews to occur 6 weeks after completion of psychoeducation program.
  Research suggests that brief, systems-focused family psychoeducation programs are useful in the treatment of Operational Stress Injuries (OSIs), specifically traumatic stress disorder (PTSD), leading to increases in targeted PTSD knowledge and skills and enhancing resilience. The purpose of this pilot study is to evaluate the perceived efficacy and utility of a pilot family psychoeducation program developed and implemented in collaboration with researchers at the Nova Scotia Health Authority (NSHA) and Mount St. Vincent University (MSVU). Using an ecological family systems theoretical framework, researchers will conduct individual semi-structured interviews with participants (based on a de novo interview guide) before, upon completion of the program, and 6 weeks after program completion to qualitatively analyze the data.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Norris, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Nova Scotia OSI Clinic, Dartmouth, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armour C, Contractor A, Elhai JD, Stringer M, Lyle G, Forbes D, Richardson JD. Identifying latent profiles of posttraumatic stress and major depression symptoms in Canadian veterans: Exploring differences across profiles in health related functioning. Psychiatry Res. 2015 Jul 30;228(1):1-7. doi: 10.1016/j.psychres.2015.03.011. Epub 2015 Apr 22. PMID 25936834
- [Background] Bowen, G. L., & Martin, J. A. (2011). The resiliency model of role performance for service members, veterans, and their families: A focus on social connections and individual assets. Journal of Human Behavior in the Social Environment, 21(2), 162-178. doi:101080/10911359.2011.546198
- [Background] Bronfenbrenner, U. (1977). Toward an experimental ecology of human development. American Psychologist, 32(7), 513-531. doi.10.1037/0003-066X.32.7.51
- [Background] Bronfenbrenner, U., & Morris, P. A. (1998). The ecology of developmental processes. In W. Damon & R. M. Lerner (Eds.), Handbook of child psychology: Theoretical models of human development (pp. 993-1028). Hoboken, NJ: John Wiley & Sons Inc
- [Background] Cramm, H., Norris, D., Smith-Evans, K., Hill, S., & Mahar, A. (2018). Military families and resiliency: Final report. Ottawa, ON: Canadian Forces Morale and Welfare Services.
- [Background] Fischer, E.P., Sherman, M.D., Han, X, & Owen, R.R. (2013). Outcomes of participation in the REACH multifamily group program for veterans with PTSD and their families. Professional Psychology, 44(3), 127-134. doi:10.1037/a0032024
- [Background] Karney, B., & Crown, J. (2007). Families under stress: An assessment of data, theory, and research on marriage and divorce in the military. Washington, DC: National Defense Research Institute.
- [Background] Lepore, S. J., & Revenson, T. A. (2006). Resilience and posttraumatic growth: Recovery, resistance, and reconfiguration. In L. G. Calhoun & R. G. Tedeschi (Eds.), Handbook of posttraumatic growth: Research and practice (pp. 24-46). New York: Psychology Press.
- [Background] Marshall, C., & Rossman, G. B. (2016). Designing qualitative research (Sixth ed.). Los Angeles, California: Sage.
- [Background] Masten AS. Global perspectives on resilience in children and youth. Child Dev. 2014 Jan-Feb;85(1):6-20. doi: 10.1111/cdev.12205. Epub 2013 Dec 16. PMID 24341286
- [Background] Monk, J.K., Ruhlman, L.M., Nelson Goff, B.S., & Ogolsky, B.G. (2018). Brief-systemic programs for promoting mental health and relationship functioning in military couples and families. Journal of Family Theory and Review, 10(3), 566-586. doi:10.1111/jftr.12280
- [Background] National Defense and The Canadian Armed Forces Ombudsman (2013). On the homefront: assessing the wellbeing of Canada's military families in the new millennium. Available from: http://www.ombudsman. forces.gc.ca/en/ombudsman-reports-stats-investigations-military-families/military-families-index.page
- [Background] Norris, D., Cramm, H., Eichler, M., Tam-Seto, L., & Smith-Evans, K. (2015). Operational stress injury: The impact on family mental health and well-being: A report to Veterans Affairs Canada. Retrieved from https://cimvhr.ca/documents/Appendix%20B.pdf?cimlang=e
- [Background] Norris, D., Cramm, H., Schwartz, K. D., Tam-Seto, L., Mahar, A. L., Eichler, M., Blackburn, D. (2018). Qualitative study on the health and well-being of families of Canadian Armed Forces veterans with mental health problems: A report to Veteran's Affairs Canada. Charlottetown, Prince Edward Island: Veterans Affairs Canada.
- [Background] Richardson JD, Contractor AA, Armour C, St Cyr K, Elhai JD, Sareen J. Predictors of long-term treatment outcome in combat and peacekeeping veterans with military-related PTSD. J Clin Psychiatry. 2014 Nov;75(11):e1299-305. doi: 10.4088/JCP.13m08796. PMID 25470095
- [Background] Richardson JD, St Cyr KC, McIntyre-Smith AM, Haslam D, Elhai JD, Sareen J. Examining the association between psychiatric illness and suicidal ideation in a sample of treatment-seeking Canadian peacekeeping and combat veterans with posttraumatic stress disorder PTSD. Can J Psychiatry. 2012 Aug;57(8):496-504. doi: 10.1177/070674371205700808. PMID 22854032
- [Background] Rosa, E. M. & Tudge, J. (2013). Urie Bronfenbrenner's theory of human development: Its evolution from ecology to bioecology. Journal of Family Theory and Review, 5, 243-258. doi:10.1111/jftr.12022
- [Background] Rutter, M. (1999). Resilience concepts and findings: Implications for family therapy. Journal of Family Therapy, 21(2), 119-144. doi:10.1111/1467-6427.00108
- [Background] Strauss, A. L., & Corbin, J. M. (1990). Basics of qualitative research: grounded theory procedures and techniques. Newbury Park, Calif: Sage.
- [Background] Thompson, J. M., Van Til, L. D., Poirier, A., Sweet, J., McKinnon, K., Sudom, K., & Pedlar, D. (2014). Health and well-being of Canadian Armed Forces Veterans: Findings from the 2013 life after service survey. Charlottetown, Prince Edward Island: Veterans Affairs Canada.
- [Background] Walsh, F. (2002). A family resilience framework: Innovative practice applications. Family Relations, 51(2), 30-137. doi:10.1111/j.1741-3729.2002.00130.x